CLINICAL TRIAL: NCT05789745
Title: Single-center, Randomized, Double-blind, Placebo-controlled, Ascending-Dose Study to Evaluate the Safety and Pharmacokinetics of Recombinant Human Plasma Gelsolin (Rhu-pGSN) After Intravenous Administration to Healthy Volunteers
Brief Title: A Study to Evaluate Plasma Gelsolin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioAegis Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTI-101
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Volunteers; Healthy
Keywords: safety; pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Doses prepared by unblinded pharmacist. Placebo and Drug are undistinguishable in syringe for administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- rhu-pGSN (Experimental): Treated with 5 doses of rhu-pGSN
  Interventions: Drug: Recombinant human plasma gelsolin
- normal saline (Placebo Comparator): Treated with 5 doses of saline
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Recombinant human plasma gelsolin — intravenous administration of either 6, 12, 18, or 24 mg/kg at time 0, 12, 36, 60 and 84 hours
  Arms: rhu-pGSN
Other: placebo — intravenous administration of saline control at time 0, 12, 36, 60 and 84 hours
  Arms: normal saline

SUMMARY:
Study BTI-101 is a Phase 1, randomized, double-blind, placebo-controlled, dose escalation, parallel design study to evaluate the safety, tolerability, and pharmacokinetics of IV rhu-pGSN or saline placebo administered as 5 doses each of 6, 12, 18, or 24 mg/kg of body weight. Each of 4 dosing cohorts will include 8 subjects randomized 3:1 rhu-pGSN:placebo (6 rhu-pGSN subjects:2 placebo subjects). Subjects will be healthy adult volunteers 18-55 years of age.

DETAILED DESCRIPTION:
Doses will be administered at 0 hours (Day 1), 12 hours (Day 1), 36 hours (Day 2), 60 hours (Day 3), and 84 hours (Day 4). Subjects will be kept in-house until after the last blood sample is taken on Day 5. Subjects will return for follow-up 7 days after the initiation of therapy (Day 8) and on Day 28 for the End-of-Study (EOS) Visit. After each cohort has completed the Day 8 visit, review of the safety results (including labs) will be conducted (and unblinded where appropriate) before the initiation of the next higher dose cohort.

To assess safety and tolerability, subjects will undergo physical examinations (including vital sign measurements), adverse event (AE) assessments, concomitant medication assessments, and safety laboratory testing. Blood samples will be collected for analysis of pGSN levels and antibodies against pGSN.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female adults 18 to 55 years of age without chronic or active acute medical conditions
2. Informed consent obtained from subject
3. Weight ≤100 kg and body mass index (BMI) <30 kg/m2
4. Willingness to use contraception during the course of the study, starting at screening and for at least 3 months after their final study treatment

Exclusion Criteria:

1. Pregnant or lactating women
2. Acute illness during the month prior to screening
3. Circumstances that may require any medications (including prescription medication, over-the-counter medication, vitamins, or supplements) during the during the inpatient days of the study other than acetaminophen
4. Hospitalization during the year prior to screening
5. History of cancer or treatment with systemic chemotherapy or radiation therapy at any time
6. Transplantation of hematopoietic or solid organs
7. History of diabetes mellitus; myocardial infarction, angina, or other cardiovascular disease; stroke or cerebrovascular disease; chronic obstructive pulmonary disease (COPD) or asthma; deep vein thrombosis (DVT)/pulmonary embolism (PE); liver or kidney disease; clinically significant psychiatric condition; or active or chronic infection
8. Receipt of blood products during the year prior to screening
9. Chronic mechanical ventilation or dialysis
10. Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results as judged by the Investigator
11. Any clinically significant abnormalities of vital signs, EKG or physical examination findings as judged by the Investigator
12. Positive results for recreational drugs during screening
13. Any other condition deemed by the Investigator as possibly interfering with the conduct of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J DiNubile, MD, Study Director — BioAegis Therapeutics
Locations (1):
- Nucleus Network, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (6 mg/kg); Cohort 2 (12 mg/kg); Cohort 3 (18 mg/kg); Cohort 4 (24 mg/kg): IV rhu-pGSN administered at 0 hours (Day 1), 12 hours (Day 1), 36 hours (Day 2), 60 hours (Day 3), and 84 hours (Day 4)
- Placebo Cohorts 1-4: Dosed at a weight-based volume of 0.025 mL/mg × dose in mg/kg × weight in kg of 0.9% saline solution via IV push (matching the volume of rhu-pGSN for a subject of that size) injected at ≤20 mL/minute though a standard 0.2 μ filter. Placebo was administered on the same schedule as the active drug.
Period: Overall Study
Arm/Group | Cohort 1 (6 mg/kg) | Cohort 2 (12 mg/kg) | Cohort 3 (18 mg/kg) | Cohort 4 (24 mg/kg) | Placebo Cohorts 1-4
Started | 6 | 6 | 6 | 6 | 8
Completed | 6 | 6 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (6 mg/kg) | Cohort 2 (12 mg/kg) | Cohort 3 (18 mg/kg) | Cohort 4 (24 mg/kg) | Placebo Cohorts 1-4 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (10.23) | 42.2 (4.07) | 37.7 (14.68) | 37.0 (15.44) | 30.5 (7.37) | 36.2 (11.00)
Age, Continuous [Median (Full Range); unit: years] | 34.0 [25 to 54] | 41.5 [38 to 48] | 36.0 [20 to 55] | 37.5 [20 to 52] | 28.5 [21 to 43] | 36.5 [20 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 3 | 1 | 12
  Male | 4 | 3 | 3 | 3 | 7 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 1 | 1 | 5
  Not Hispanic or Latino | 4 | 5 | 6 | 5 | 7 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 3 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2 | 4
  White | 5 | 5 | 5 | 3 | 6 | 24
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.55 (2.899) | 24.77 (3.506) | 25.28 (3.722) | 25.43 (2.876) | 23.85 (2.021) | 24.72 (2.862)
BMI [Median (Full Range); unit: kg/m^2] | 24.50 [19.5 to 27.9] | 24.65 [20.8 to 28.8] | 26.60 [19.0 to 29.7] | 25.95 [21.9 to 29.1] | 23.85 [21.2 to 26.4] | 24.75 [19.0 to 29.7]

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of subjects who had an Adverse Event
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (6 mg/kg) | Cohort 2 (12 mg/kg) | Cohort 3 (18 mg/kg) | Cohort 4 (24 mg/kg) | Placebo Cohorts 1-4
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Participants | 1 | 2 | 3 | 2 | 1

2. Primary Outcome: Serious Adverse Events
Description: Number of subjects who had a Serious Adverse Event
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (6 mg/kg) | Cohort 2 (12 mg/kg) | Cohort 3 (18 mg/kg) | Cohort 4 (24 mg/kg) | Placebo Cohorts 1-4
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Participants | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Pharmacokinetics: pGSN Concentration
Description: Concentration of pGSN at baseline, 12 hours after dose 1, and 24 hours after doses 2 and 5
Time Frame: 108 hours
Measure: Geometric Mean (Standard Deviation); unit: micrograms/mL
Arm/Group | Cohort 1 (6 mg/kg) | Cohort 2 (12 mg/kg) | Cohort 3 (18 mg/kg) | Cohort 4 (24 mg/kg)
Number analyzed (Participants) | 6 | 6 | 5 | 6
micrograms/mL
  Baseline | 63.6 (13.2) | 61.2 (19.7) | 59.1 (8.8) | 71.8 (11.1)
  Cmax (Dose 1) | 148.4 (26.8) | 347.5 (41.2) | 442.5 (50.2) | 663.6 (110.8)
  Cmax (Dose 2) | 225.2 (27.0) | 506.9 (78.5) | 691.5 (110.5) | 855.7 (200.6)
  Cmax (Dose 5) | 218.9 (37.7) | 501.6 (60.4) | 703.8 (140.7) | 970.9 (87.9)

4. Secondary Outcome: Pharmacokinetics: pGSN Area Under the Curve (AUC)
Description: Area Under the Curve (AUC) of pGSN concentration at 12 hours after dose 1, and 24 hours after doses 2 and 5
Time Frame: 108 hours
Measure: Geometric Mean (Standard Deviation); unit: hours*(micrograms/mL)
Arm/Group | Cohort 1 (6 mg/kg) | Cohort 2 (12 mg/kg) | Cohort 3 (18 mg/kg) | Cohort 4 (24 mg/kg)
Number analyzed (Participants) | 6 | 6 | 5 | 6
hours*(micrograms/mL)
  AUC0-12 (dose 1) | 1245.5 (257.9) | 2737.5 (379.1) | 3547.0 (657.3) | 4832.3 (646.6)
  AUC0-24 (dose 2) | 3066.2 (256.8) | 6448.5 (599.5) | 9374.2 (2456.0) | 10258.2 (2035.6)
  AUC0-24 (dose 5) | 3486.5 (1035.2) | 6599.1 (1334.2) | 9139.1 (793.1) | 12135.3 (1172.4)

5. Secondary Outcome: Pharmacokinetics: pGSN Half-life
Description: Half-life of pGSN concentration 12 hours after dose 1, and 24 hours after doses 2 and 5
Time Frame: 108 hours
Measure: Geometric Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 (6 mg/kg) | Cohort 2 (12 mg/kg) | Cohort 3 (18 mg/kg) | Cohort 4 (24 mg/kg)
Number analyzed (Participants) | 6 | 6 | 5 | 6
hours
  t1/2 (dose 1) | 14.0 (5.4) | 13.1 (2.6) | 9.2 (3.0) | 10.7 (5.2)
  t1/2 (dose 2) | 16.7 (6.1) | 14.5 (3.4) | 15.1 (4.5) | 12.0 (1.5)
  t1/2 (dose 5) | 28.4 (8.5) | 22.0 (11.3) | 17.6 (1.9) | 14.5 (2.2)

6. Secondary Outcome: Presence of Anti-drug Antibodies
Description: Number of participants who tested positive for anti-pGSN antibodies at baseline, and on day 28
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (6 mg/kg) | Cohort 2 (12 mg/kg) | Cohort 3 (18 mg/kg) | Cohort 4 (24 mg/kg) | Placebo Cohorts 1-4
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Participants
  Baseline | 0 | 0 | 0 | 0 | 0
  Day 28 | 0 | 0 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: From the first study intervention to 4 weeks
Arm/Group | Cohort 1 (6 mg/kg) | Cohort 2 (12 mg/kg) | Cohort 3 (18 mg/kg) | Cohort 4 (24 mg/kg) | Placebo Cohorts 1-4
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 1/6 | 2/6 | 3/6 | 2/6 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (6 mg/kg) (N=6) | Cohort 2 (12 mg/kg) (N=6) | Cohort 3 (18 mg/kg) (N=6) | Cohort 4 (24 mg/kg) (N=6) | Placebo Cohorts 1-4 (N=8)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Muscle contractions involuntary (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT05789745/Prot_SAP_000.pdf